CLINICAL TRIAL: NCT01431404
Title: Randomized,Double-blind,Single-dosing,Crossover Study to Compare the Safety and Pharmacokinetic Characteristics of HD203 With Active Comparator
Brief Title: Safety and Pharmacokinetic Characteristics of HD203 Liq. in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanwha Chemical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAGLE-I-11
Record Dates: First submitted 2011-09-05; First posted 2011-09-09 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enbrel, prefilled syringe (Active Comparator)
  Interventions: Biological: Etanercept (Enbrel)
- HD203, prefilled syringe (Experimental)
  Interventions: Biological: HD203

INTERVENTIONS:
Biological: Etanercept (Enbrel) — prefilled syringe, SC
  Arms: Enbrel, prefilled syringe
Biological: HD203 — HD203, prefilled syringe, SC injection
  Arms: HD203, prefilled syringe

SUMMARY:
The purpose of this study is compare the safety and pharmacokinetic characteristics of HD203 liquid with those of etanercept (enbrel) prefilled injection after subcutaneous injection.

DETAILED DESCRIPTION:
A randomized, double-blind, single-dosing, crossover study to compare the safety and pharmacokinetic characteristics of HD203 Liquid 25 mg with those of Enbrel Prefilled® injection 25 mg after subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years of healthy volunteers
* Weight over 55kg
* Subject who signed on ICF

Exclusion Criteria:

* Subject who had been treated with Etanercept before

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | up to 49days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea